CLINICAL TRIAL: NCT06179173
Title: Is High-intensity Aerobic Interval Training Appropriate for Recovering Impairments and Activity Limitations in the Acute Phase of Stroke? A Randomized Controlled Trial in Benin
Brief Title: Effectiveness of High-intensity Aerobic Interval Training on Impairments and Activity Limitations in the Acute Phase of Stroke in Benin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: Université de Parakou (Other)
Responsible Party: Principal Investigator, Dominique Hansen, Full Professor of Rehabilitation and Exercise Physiology in Cardiometabolic Diseases, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLERB-UP023/2023
Record Dates: First submitted 2023-10-03; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT-RCE (Experimental): All participants will receive conventional physiotherapy for half an hour thrice weekly for six weeks. Conventional physiotherapy will be followed by a 15 min rest period, then the HIIT on a semi-recumbent cycle SOLE R92 (HIIT-RCE) will be performed.Each HIIT-RCE session will be preceded by 3-min of unloaded cycling as a warm-up and ended with 3-min of stretching. The HIIT-RCE procedure will start at 4-min at 30% of the peak workload interspersed with 1-min at 70% of the peak workload for weeks 1-2 (4 repetitions for 20 min) and increased by approximately 5 minutes every two weeks as tolerated to reach 30 minutes from week 5 (6 repetitions). The training intensity will progress similarly by 5% peak work rate two weeks as tolerated to reach 4-min at 40% peak workload interspersed with 1-min 80% peak workload from week-5. The cycle frequency will be at least 50 rpm.
  Interventions: Other: HIIT-RCE
- Conventional physiotherapy (Active Comparator): The group will receive conventional physiotherapy that will consist primarily of passive movement, stretching, balance training, strengthening, and lower intensity overground walking for 30 minutes. This will be followed by a 15-minute rest period. Then an unloaded cycling session on a semi-recumbent cycle ergometer with preferred cadence until to get equal energy expenditure per session between groups by case-matching.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Other: HIIT-RCE — High-intensity interval training on semi-recumbent cycle ergometer
  Arms: HIIT-RCE
Other: Conventional physiotherapy — Conventional physiotherapy
  Arms: Conventional physiotherapy

SUMMARY:
This clinical trial aims to examine the effects of combining HIIT on a semi-recumbent cycle ergometer (HIIT-RCE) with conventional physiotherapy on impairments and activity limitations in early subacute stroke. We hypothesized that HIIT combined with conventional physiotherapy would be more effective than conventional physiotherapy in improving workload capacity.

ELIGIBILITY:
Inclusion Criteria:

People with the diagnosis of stroke were screened and recruited within the first-month after the stroke onset according to the following criteria

1. first episode from an ischemic or hemorrhagic stroke confirmed by CT scan;
2. muscle strength of the affected leg defined by Motricity Index between 14 and 19, i.e., between 2 and 4 on the Medical Research Council scale;
3. modified Ashworth score of 0 or 1, indicating no spasticity or slight spasticity over the affected lower limb, respectively
4. able to walk at least 5 meters independently with or without assistive devices and understand simple instructions;
5. resident in Parakou or its surroundings
6. wish to participate in the hospital program

Exclusion Criteria:

Patients whose medical records reported

1. uncontrolled cardiac arrhythmias (e.g. atrial fibrillation, ventricular tachycardia), heart failure, or recent myocardial infarction, arteriopathy,
2. primary orthopedic conditions (e.g., fractures, active rheumatoid arthritis),
3. other neurological diseases (such as Parkinson's disease and Alzheimer's disease), (4) patients unable to perform a graded exercise test, i.e., unable to reach the target cadence of 50 rpm or exercise-induced asthma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Workload capacity | At enrolment (T0), After 6 weeks of intervention (T1), 3 months (T2) and 6 months (T3) after intervention
  A progressive intensity maximal effort cycling test will be performed in a semi-recumbent ergometer cycle (SOLE R90) to determine each participant's peak workload (in watts).

SECONDARY OUTCOMES:
The Berg Balance Scale (BBS), | At enrolment (T0), After 6 weeks of intervention (T1), 3 months (T2) and 6 months (T3) after intervention
  The BBS will be used to assess balance impairment. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. The minimum score is 0 and the maximum score is 56. A score of 56 indicates functional balance and a score < 45 indicates a higher risk of falling.
The 6-minute walk test (6MWT) | At enrolment (T0), After 6 weeks of intervention (T1), 3 months (T2) and 6 months (T3) after intervention
  The 6MWT is a measure of walking endurance. 35,36 It assesses the distance a participant can walk as fast as possible for 6 min on a 30 m straight line with the option to stop for fatigue at any point.
The 10-meter Walk Test (10mWT) | At enrolment (T0), After 6 weeks of intervention (T1), 3 months (T2) and 6 months (T3) after intervention
  The 10mWT is a performance measure used to assess walking speed in meters per second over the middle 10 meters of a 14-meter course.
The 5-Repetition Sit-To-Stand test (5R-STS) | At enrolment (T0), After 6 weeks of intervention (T1), 3 months (T2) and 6 months (T3) after intervention
  The 5R-STS test measures the time to complete five repetitions of the sit-to-stand maneuver. Participants unable to complete five repetitions within 1-min will be given a score of 60 s.
The EQ-5D-5L | At enrolment (T0), After 6 weeks of intervention (T1), 3 months (T2) and 6 months(T3) after intervention
  The EQ-5D-5L is a self-assessed, health-related, quality of life questionnaire validated for acute stroke. It has 5 domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) of 5 items each, and scores range from 0 (best quality of life) to 1 (worst quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Dominique R Hansen, PhD, Principal Investigator — Hasselt University
Locations (1):
- University Hospital of Parakou, Parakou, Benin

IPD SHARING:
Plan to Share IPD: No
Data will be available to researchers upon request to the first author (ERA)

REFERENCES:
- [Derived] Amanzonwe ER, Noukpo SI, Adoukonou T, Bonnechere B, Feys P, Hansen D, Kossi O. Exercise Intensity Matters in the Rehabilitation of Stroke in the Acute Stage: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2025 Nov;39(11):892-905. doi: 10.1177/15459683251356969. Epub 2025 Aug 11. PMID 40788139